CLINICAL TRIAL: NCT03601780
Title: Effect of Local Wound Infiltration Plus Usual Care Versus Usual Care Alone on Pain Relief After Open Renal Surgery.
Brief Title: Local Wound Infiltration in Renal Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM62018
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local wound infiltration (Active Comparator): local wound infiltration plus usual care
  Interventions: Drug: local wound infiltration plus usual care
- Control (Placebo Comparator): usual care only
  Interventions: Drug: usual care only

INTERVENTIONS:
Drug: local wound infiltration plus usual care — local wound infiltration plus usual care
  Arms: Local wound infiltration
Drug: usual care only — usual care only
  Arms: Control

SUMMARY:
Multimodal analgesia is a rational approach to treat various components of postoperative pain.

DETAILED DESCRIPTION:
Local anesthetic wound infiltration is widely recognized as a useful adjunct during multimodal postoperative pain management whether given before operation or perioperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II, aged between 30 and 65 yr, and undergoing open renal surgery

Exclusion Criteria:

* history of adverse reactions to local anaesthetics, chronic hepatic disease, chronic renal disease chronic pain, chronic preoperative opioid consumption, psychiatric disorders which would prevent postoperative assessments,

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | The first 48 hours after surgery
  Visual analogue scale ranging from 0-10 cm where 0 cm
  = no pain and 10 cm = the worst imaginable pain.